CLINICAL TRIAL: NCT02723253
Title: Concurrent Chemoradiation With Concomitant Boost In Locally Advanced Rectal Cancer: A Phase II Study.
Brief Title: Concurrent Chemoradiation With Concomitant Boost In Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Associate Professor of Gastroenterology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOMOX Rectal Study
Record Dates: First submitted 2016-03-19; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; radiotherapy; chemotherapy; Raltitrexed; Oxaliplatin
MeSH Terms: conditions — Rectal Neoplasms | interventions — Radiotherapy; raltitrexed; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy plus Tom-Ox (Experimental): Patients received concomitant boost RT (55 Gy/5 weeks) with concurrent Tom-Ox chemotherapy. The concurrent chemotherapy consisted of 15 min intravenous infusion Raltitrexed (Tomudex ®) 3 mg/m2 and a two-hours intravenous infusion of Oxaliplatin (Eloxatin ®) at 130 mg/m 2, 20 min after raltitrexed, on days 1, 17, 35.
  Interventions: Radiation: Radiotherapy; Drug: Tom-OX

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy was applied as conformal 3-D technique and was delivered with photon energies of 10 - 15 MV. The beams were delivered by an Elekta Precise Linac equipped with standard multi leaf collimators (MLC). A daily online check of isocenter position was performed using portal imaging, with set-up correction in case of displacement > 0.5 cm in any direction. Radiation dose delivered to PTV2 was 45 Gy (1.8 Gy/fraction) with a concomitant boost dose to the PTV1 of 10 Gy with accelerated fractionation at 2.2 Gy/fraction, five consecutive days for week.
Drug: Tom-OX — The concurrent chemotherapy consisted of 15 min intravenous infusion Raltitrexed (Tomudex ®) 3 mg/m2 and a two-hours intravenous infusion of Oxaliplatin (Eloxatin ®) at 130 mg/m 2, 20 min after raltitrexed, on days 1, 17, 35.
  Other Names: Tomudex ®, Eloxatin ®

SUMMARY:
Neoadjuvant chemoradiation (CRT), is considered the standard treatment of locally advanced rectal cancer with a positive impact on locoregional control and survival.However, patients with T4 rectal cancer show high risk of local recurrence after conventional treatment. Therefore investigators designed a prospective Phase II study on patients with locally advanced rectal cancer or locally recurrences, to evaluate the efficacy in terms of pathological response and resectability of concomitant boost RT (55 Gy/5 weeks) with concurrent Raltitrexed and Oxaliplatin (Tom-Ox) chemotherapy.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiation (CRT), is considered the standard treatment of locally advanced rectal cancer with a positive impact on locoregional control and survival. However, patients with T4 rectal cancer show high risk of local recurrence (LR) after conventional treatment. This was a prospective Phase II study on patients with locally advanced rectal cancer or locally recurrences, to evaluate the efficacy in terms of pathological response and resectability of concomitant boost RT (55 Gy/5 weeks) with concurrent Raltitrexed and Oxaliplatin (Tom-Ox) chemotherapy. The primary aim was to assess the pathological complete response rate. Key secondary aim was the resectability. Secondary aims were evaluation of treatment-related acute and late toxicity, local control, disease-free survival and overall survival (OS). The follow-up period of each subjects started after the radiochemotherapy treatment and ended after a maximum of 36 months of observation or until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced (T4N0-2) or locally recurrent rectal adenocarcinoma;
* Age ≥ 18 years;
* Eastern Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

* Metastatic patients
* unfit surgery patients,
* pregnant or breast feeding females
* patients with clinically detectable ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of patients defined as good responders (G1 or G2) according to the Mandard regression grading system. | 8 weeks after chemo-radiotherapy
  Pathologic responses of the primary tumours were defined according to the Mandard regression grading system: grade 1 was recorded when no tumour cells remained in the primary tumour and lymph nodes (pCR); grade 2 was characterized by the presence of rare residual cancer cells scattered through the fibrosis; grade 3 was characterized by an increase in the number of residual cancer cells, but fibrosis still predominated; grade 4 showed residual cancer outgrowing fibrosis; and grade 5 was characterized by an absence of regressive changes. Good responders were defined those patients with a pathologic response with Mandard G1 or G2 and poor responder patients with Mandard G3, G4 or G5.

SECONDARY OUTCOMES:
Number of patients in which a surgical resection was feasible | 8 weeks after chemo-radiotherapy
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | Up to 36 months. In details, follow-up examinations were performed 4 weeks after surgery and every 6 months until the established length of follow-up or death.
  CTCAE v 3.0 was used to score acute and late radiation toxicity.
The number of patients without disease (i.e. rectal cancer) during the follow-up. | Up to 36 months.
  The disease-free survival (DFS) was defined as the time from the diagnosis to the documented local or distant recurrence or last follow-up.
The number of patients still alive at the end of follow-up | Up to 36 months
  The overall-survival (OS) was defined as the time from the diagnosis until death for any cause or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, Prof, Study Director — Division of Radiation Oncology, S.Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No